CLINICAL TRIAL: NCT06886321
Title: Evaluation of the Effectiveness of Irreversible Electroporation for the Treatment of Prostate Cancer
Brief Title: Prostate Irreversible Electroporation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Hang Yee, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2023.215
Record Dates: First submitted 2025-03-05; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Focal therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Prostate Irreversible Electroporation (Experimental)
  Interventions: Device: Prostate Irreversible Electroporation

INTERVENTIONS:
Device: Prostate Irreversible Electroporation — The Prostate Irreversible Electroporation procedure was performed in our institution by a single urologist using an Prostate Irreversible Electroporation device and 18-gauge electrodes (Nanoknife®; Angiodynamics, Queensbury, NY, USA). All patients were positioned in lithotomy position under general anesthesia. A transrectal ultrasound was used to visualize the prostate and a brachytherapy grid was used to place the electrodes. An indwelling catheter was placed to empty the bladder. Four to six electrodes were placed through the perineum via the template grid to surround the targeted lesion. The lesion was defined based on prostate biopsy and MRI images. The active tip varied between 15- and 20-mm exposure. The distances between the electrodes were measured using TRUS and entered into the Nanoknife system. An initial ten pulses were delivered to ensure sufficient current was delivered between the electrodes (20-40 A). If sufficient then the remaining 80 pulses were given.

SUMMARY:
Conventional treatment options for localized prostate cancer include prostatectomy, radiotherapy and active surveillance. However, prostatectomy and radiotherapy carry certain degree of morbidity, including the risks of urinary incontinence, erectile dysfunction and injury to the structures in the proximity. Active surveillance carries the risk of disease progression and psychological distress to the patients. Focal therapy employs the concept of only destroying the significant lesion, resulting in disease cure and improved functional outcome. Among the different options of focal therapy, Irreversible electroporation has evolved over the past decades and can be a reliable treatment option. Our study aims at assess the safety and effectiveness of such treatment in prostate cancer management.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 40 - 85 years
* Visible index lesion(s) on MRI
* Found to have localized prostate cancer after MRI-USG fusion targeted biopsy or USG-guided template biopsy: Clinical tumour stage <=T2, or Gleason score <=7, or PSA <= 20 ng/ml

Exclusion Criteria:

* Patients unfit for contrast MRI exam
* Patients with active urinary tract infection
* Patients with bladder pathology including bladder stone and bladder cancer
* Patients with urethral stricture
* Patients with neurogenic bladder and/or sphincter abnormalities
* Patients who fail to give informed consent

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
6-month oncological outcome | 6-month after treatment
  6-month oncological outcome after Prostate Irreversible Electroporation treatment, as defined by multiparametric MRI result of prostate

SECONDARY OUTCOMES:
6-month and 12-month functional and oncological outcome | At 6-month and 12-month after treatment
  6-month and 12-month functional and oncological outcome after Prostate Irreversible Electroporation treatment by questionnaires and multiparametric MRI result of prostate
30-day complications | at 30 day after treatment
  30-day complications after study intervention
Presence of histologically proven prostate cancer recurrence | At 12-month after treatment
  Presence of histologically proven prostate cancer recurrence on biopsy in suspicious cases
PSA change | At 3-month, 6-month, 9-month and 12-month after treatment
  PSA change after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hang Yee, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No